CLINICAL TRIAL: NCT04385992
Title: A Prospective Phase II Single-Arm Trial on Neoadjuvant Peptide Receptor Radionuclide Therapy With 177Lu-DOTATATE Followed by Surgery for Resectable Pancreatic Neuroendocrine Tumors
Brief Title: Neoadjuvant PRRT With 177Lu-DOTATATE Followed by Surgery for Resectable PanNET
Acronym: NeoLuPaNET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Massimo Falconi, Professor, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neo.Lu.Pa.NET
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All enrolled patients (Experimental): Enrolled patients following inclusion criteria
  Interventions: Drug: 177Lu-Dotatate

INTERVENTIONS:
Drug: 177Lu-Dotatate — Peptide Receptor Radionuclide Therapy (PRRT) is based on specific somatostatin receptor targeting with radiolabelled analogues 90Y-DOTATOC and 177Lu-DOTATATE

SUMMARY:
Peptide Receptor Radionuclide Therapy (PRRT) is based on specific somatostatin receptor targeting with radiolabelled analogues 90Y-DOTATOC and 177Lu-DOTATATE. These two most commonly used radiopeptides, 90Y-DOTATOC and 177Lu-DOTATATE, produce overall objective response rates of 15-35%. PRRT is generally well tolerated with mild toxicity, if the necessary precautions, such as the co-administration of nephroprotective amino acids or the adjustment of the administered activity, are taken.

The main aim of this study is to evaluate the safety and the efficacy of neoadjuvant PRRT with 177Lu-DOTATATE followed by surgical resection for resectable non-functioning PanNETs at high risk of recurrence.

The primary endpoint is the Rate of postoperative 90-day morbidity and mortality after neoadjuvant PRRT with 177Lu-DOTATATE followed by pancreatic resection and the secondary endpoints are:

1. Rate of objective radiological response to PRRT with 177Lu-DOTATATE according to RECIST criteria (version 1.1), for primary lesions' assessment, and modified RECIST criteria (mRECIST), for liver metastases' assessment, if detected
2. Quality of life (QoL) after neoadjuvant PRRT followed by pancreatic surgical resection.

The study is designed as a prospective phase II single-arm trial. 8 Italian centers will participate to the study (6 surgical sites, 2 nuclear medicine sites).

Patients will be recruited for 12 months. The study will end 2 months after operation of the last patient enrolled and the total duration of the study will be 24 months.

Sample size estimation: 30 patients

DETAILED DESCRIPTION:
Rationale:

In a recent study un initial experience was reported with neoadjuvant PRRT followed by surgical resection in patients affected by PanNETs. In this study, patients with resectable or potentially resectable PanNETs at high risk of recurrence after surgery who underwent neoadjuvant PRRT were compared with a group of patients who underwent upfront surgery. Of note, patients who underwent neoadjuvant PRRT had a significant lower risk of developing pancreatic fistula and a lower risk of postoperative complications. Moreover, among those patients who underwent curative resection, patients who received PRRT had a progression-free survival significantly longer after compared to upfront surgery. Neoadjuvant PRRT may be a valuable option to reduce the risk of failure after surgery in patients with PanNETs who are at high risk of recurrence. Nevertheless, the safety and the efficacy of neoadjuvant PRRT has never been investigated in a prospective trial.

The main aim of this study is to evaluate the safety and the efficacy of neoadjuvant PRRT with 177Lu-DOTATATE followed by surgical resection for resectable non-functioning PanNETs at high risk of recurrence.

The primary endpoint is the Rate of postoperative 90-day morbidity and mortality after neoadjuvant PRRT with 177Lu-DOTATATE followed by pancreatic resection and the secondary endpoints are:

1. Rate of objective radiological response to PRRT with 177Lu-DOTATATE according to RECIST criteria (version 1.1), for primary lesions' assessment, and modified RECIST criteria (mRECIST), for liver metastases' assessment, if detected.
2. Quality of life (QoL) after neoadjuvant PRRT followed by pancreatic surgical resection.

The study is designed as a prospective phase II single-arm trial. 8 Italian centers will participate to the study (6 surgical sites, 2 nuclear medicine sites).

Patients will be recruited for 12 months. The study will end 2 months after operation of the last patient enrolled and the total duration of the study will be 24 months.

Sample size:

By using the Single-Stage Phase II sample size method, we estimated a sample size of 30 patients to test if the proportion of patients without postoperative complications (responses) is more than or equal to 57% (p1 ) or less than equal to 39% (p0 ).

To be enrol in the study, all the patients should have a cytological/histological confirmation of PanNET and meet one or more inclusion criteria. Moreover, all the exclusion criteria should have been ruled out.

Patients will undergo the following laboratory examinations at week 0, week 1, week 9, week 17, week 25, week 38, week 40, week 45-52: blood cell count, urea, creatinine, sodium, potassium, cloride, calcium, glucose, bilirubin, AST, ALT, LDH, GGT, ALP, Albumin, urine test. Gravindex will be executed at week 0, week 1, week 9, week 17, week 25, week 40 and they will be asked to fill a quality of life questionnaire at wwk 0, week 38, week 40-52.

Enrolled patients will be treated with standard pancreatic resection according to PanNET localization, after a course (4 cycles) of neoadjuvant PRRT with 177Lu-DOTATATE.

Patients will receive a cumulative activity of 29.600 MBq (800 mCi), divided in 4 administrations (or cycles) of 7.400 MBq (200 mCi) each, with treatment intervals of 6-8 weeks. The per-cycle activity of 177Lu-DOTATATE (and consequently the cumulative activity) might be reduced if relevant blood and renal toxicity, or other side effects, will occur during the course of PRRT.

177Lu-DOTATATE will be slowly injected intravenously over a period of 30 minutes and using a dedicated pump-system of infusion.

During the administration of the therapy, performed into a dedicated room of the Nuclear Medicine Division, the Health Physics staff will monitor the patient by means of an ionization chamber, in order to check the completeness of the radiopeptide administration.

In order to obtain an adequate hydration of the patient and to protect the renal parenchyma during the phase of excretion of the radiopharmaceutical from an excessive tubular reuptake of radiopetide, the administration of the radiopharmaceutical will be preceded and followed (without interruption) with intravenous infusion of 1000 ml of 0.9% sodium chloride solution containing L-Arginine hydrochloride and/or Lysine.

The gamma emission of 177Lu (113 and 208 KeV, relative abundance 6 and 11%, respectively) allows a suitable observation of the radiopharmaceutical biodistribution during the entire therapeutic phase.

After 16-24 hours from administration of 177Lu-DOTATATE (and for each treatment cycle) patients will undergo anterior and posterior whole body scan (imaging will be acquired on a 128x512 matrix, by means a double-headed gamma-camera, equipped with a low-energy high-resolution collimator (LEHR), with energetic window set on 177Lu peaks.) in order to verify the correct bio-distribution of the radiopharmaceutical and its focal uptake into the target lesions.

Moreover, at 1st and 4th cycle, when feasible and indicated, a more accurate imaging evaluation will be performed by using SPECT or SPECT/CT imaging (6-24 hours after administration), in order to quantify percentage of radiopharmaceutical uptake and half-life, absorbed dose, effective biological dose (BED), equivalent uniform dose (EUD) both in target lesions and critical organs (bone marrow and kidney) and correlate these parameters with the response to the treatment) and with the toxicity profile.

All patients will be re-evaluated 3 months after the 4th cycle of PRRT, in order to assess the rate of objective radiological response, according to RECIST criteria (version 1.1).

Patients will undergo standard pancreatic surgery plus lymphadenectomy at one of the participating surgical site identified in the protocol. Pancreatic resection will be performed according to the localization and extended to nearby organs and/or vessels when invasion is present. Concomitant liver resection may be performed in the presence of liver metastasis.

Assessment of outcomes. 90-day post-operative mortality and morbidity will be classified according to the definition proposed by Dindo et al.

The rate of objective radiological response to PRRT with 177Lu-OTATATE according to RECIST criteria (version 1.1), for primary lesions' assessment, and modified RECIST criteria (mRECIST), for liver metastases' assessment, if detected.

The quality of life (QoL) at diagnostic workup, after neoadjuvant PRRT and after the pancreatic surgical resection, will be evaluated by EORTC-QLQ-C30 questionnaire.

Data will be collected with CRFs and information will be recorded in a protected database.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Morphological confirmation by high-quality imaging technique (MR or CT scan)
* Cytological or histologically confirmed sporadic resectable nonfunctioning PanNETs (NF-PanNETs) with positive 68Ga-DOTATOC PET/CT (with primary lesion uptake greater than the normal liver and SUV bw max ≥ 15) and at least one of the following high-risk features:
* Radiological tumour size > 40 mm
* Well differentiated G2 NF-PanNETs with Ki67 >10% or well differentiated NF-PanNETs G3
* Presence of nearby organs involvement
* Vascular invasion (excluding the presence of superior mesenteric vein/portal vein invasion > 180° and/or celiac trunk/superior mesenteric artery invasion)
* Mesenteric and/or portal and/or splenic vein thrombosis
* Presence of a single resectable liver metastasis
* Presence of enlarged hypervascularized lymph nodes at imaging that are positive at 68Ga-DOTATOC PET/CT
* Absence of extra-abdominal disease
* Absence of peritoneal carcinomatosis
* Karnofsky Performance Status ≥ 90 or o ECOG-PS=0
* ASA ≤ 3
* Preserved hematologic, hepatic and renal parameters (WBC> 2,500/ml [ANC> 1,500/mcl]; Hb> 10g/dL; PTL> 100,000/mcl; bilirubin< 2.5 mg/dl, creatinine< 2 mg/dl)
* Absence of serious disease which can compromise safety (cardiac failure, previous myocardial infarction within prior 6 months, history of psychiatric disabilities, synchronous malignancy)

Exclusion Criteria:

* Age < 18 years
* Negative functional Imaging (68Ga-DOTATOC PET/CT)
* Presence of genetic syndrome (MEN1, VHL, NF)
* Functioning PanNET
* NF-PanNEC G3
* Absence of "high-risk features" as defined above
* Presence of extra abdominal disease
* Presence of multiple liver metastases
* Presence of peritoneal carcinomatosis
* Previous PanNET-directed treatment
* Karnofsky Performance Status < 90% or ECOG-PS > 0
* ASA > 3
* Inadequate bone marrow, liver and kidney function
* Presence of serious disease which can compromise safety (cardiac failure, previous myocardial infarction within prior 6 months, history of psychiatric disabilities, synchronous malignancy)
* Bone marrow invasion
* Life expectancy less than 6 months
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study or 5 half-life of the experimental drug
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Creatinine clearance < 30 mL/min calculated by the Cockroft Gault method
* Uncontrolled congestive heart failure (NYHA III, IV).
* Total bilirubin > 3 x normal rate
* Serum albumin < 3.0 g/dL u
* Hb concentration < 5.0 mmol/L (<8.0 g/dL); WBC < 2x10E9/L (2000/mm3); platelets < 75x10E9/L (75x10E3/mm3)
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity | from week 40 until week 52
  Rate of postoperative 90-day morbidity after neoadjuvant PRRT with 177Lu-DOTATATE followed by pancreatic resection
Postoperative mortality | from week 40 until week 52
  Rate of postoperative 90-day mortality after neoadjuvant PRRT with 177Lu-DOTATATE followed by pancreatic resection

SECONDARY OUTCOMES:
Radiological response | week 38
  Rate of objective radiological response to PRRT with 177Lu-DOTATATE according to RECIST criteria (version 1.1) and modified RECIST criteria (mRECIST), when required

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Falconi, Professor, Principal Investigator — Ospedale San Raffaele IRCCS
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No